CLINICAL TRIAL: NCT04921111
Title: A Randomized, Double-Blind, Controlled (Positive and Placebo) Phase I Clinical Trial to Estimate Safty and Immunogenicity of the SCT1000 in Healthy Women Aged 18 to 45 Years
Brief Title: A Phase I Safty and Immunogenicity Study of SCT1000 in Healthy Women Aged 18 to 45 Years
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SCT1000-01
Record Dates: First submitted 2021-05-31; First posted 2021-06-10 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: HPV Infection Vaccine Safety SCT1000
MeSH Terms: interventions — aluminum phosphate; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Women Aged 18 to 26 Years (Experimental): 120 healthy women aged18 to 26 years are in this arm. The first group was 40 subjects to be inoculated with low dose vaccine; After the first low dose group was completed, the safety observation was conducted 7 days after the first dose was completed. If there was no need to suspend / terminate the study, 40 subjects in the group were continued to receive the medium dose vaccine; After the first dose group was completed, the safety observation was 7 days after the first dose was completed. If there was no need to suspend / terminate the test, 40 subjects in the group were inoculated with high dose group. In each dose group SCT1000 : Gardasil®9 : placebo =3:1:1.
  Interventions: Drug: SCT1000; Drug: Gardasil®9; Drug: placebo
- Healthy Women Aged 27 to 45 Years (Experimental): 120 healthy women aged 27 to 45 years are in this arm. The first group was 40 subjects to be inoculated with low dose vaccine; After the first low dose group was completed, the safety observation was conducted 7 days after the first dose was completed. If there was no need to suspend / terminate the study, 40 subjects in the group were continued to receive the medium dose vaccine; After the first dose group was completed, the safety observation was 7 days after the first dose was completed. If there was no need to suspend / terminate the test, 40 subjects in the group were inoculated with high dose group. In each dose group SCT1000 : Gardasil® : placebo =3:1:1.
  Interventions: Drug: SCT1000; Drug: placebo; Drug: Gardasil®

INTERVENTIONS:
Drug: SCT1000 — Recombinant 14 valent human papillomavirus vaccine (6,11,16,18,31,33,35,39,45,51,52,56,58,59) (insect cells)
  Other Names: Recombinant 14 valent Human Papillomavirus Vaccine
Drug: Gardasil®9 — Recombinant 9 or 4 valent human papillomavirus vaccine
  Other Names: Recombinant 9 valent human papillomavirus vaccine
  Arms: Healthy Women Aged 18 to 26 Years
Drug: placebo — aluminium phosphate
  Other Names: aluminium phosphate
Drug: Gardasil® — Recombinant 4 valent human papillomavirus vaccine
  Other Names: Recombinant 4 valent human papillomavirus vaccine
  Arms: Healthy Women Aged 27 to 45 Years

SUMMARY:
A phase 1 random, double blind, positive and placebo control trail was conducted in 120 healthy women in the arm A: 18-26 years old and Arm B: 27-45 years old. The 40 subjects to be inoculated with low, middle, and high dose vaccinefirst in sequence if there was no safety issue. In each dose group SCT1000 : placebo: positive =3:1:1.Two arms can be recruited at the same time. If the DSMB assessment shows that the adverse events of a certain dose group meet the criteria of suspension / termination, the dose group will be suspended / terminated, and the vaccination of this dose group or higher dose group will not be carried out, and the study of other dose groups will continue. If this happens at a low dose, the study will be suspended / terminated.

DETAILED DESCRIPTION:
Arm A: 18-26 years old. Random, double blind, Gardasil®9 positive control and placebo control was conducted in 120 healthy women in the arm. The first group was 40 subjects to be inoculated with low dose vaccine; After the first low dose group was completed, the safety observation was conducted 7 days after the first dose was completed. If there was no need to suspend / terminate the study, 40 subjects in the group were continued to receive the medium dose vaccine; After the first dose group was completed, the safety observation was 7 days after the first dose was completed. If there was no need to suspend / terminate the test, 40 subjects in the group were inoculated with high dose group. In each dose group SCT1000 : placebo: Gardasil® 9=3:1:1.Arm B: 27-45 years old. Random, double blind, Gardasil® positive control and placebo control was conducted in 120 healthy women in the arm. The first group was 40 subjects to be inoculated with low dose vaccine; After the first dose of the low dose group was completed, the safety observation was conducted 7 days after the first dose was completed. If there was no need to suspend / terminate the study, 40 subjects in the group were continued to be inoculated in the medium dose vaccine; After the first dose group was completed, the safety observation was 7 days after the first dose was completed. If there was no need to suspend / terminate the test, 40 subjects in the group were inoculated with high dose group. SCT1000 in each dose group: placebo: Gardasil® =3:1:1.Two arms can be recruited at the same time. If the DSMB assessment shows that the adverse events of a certain dose group meet the criteria of suspension / termination, the dose group will be suspended / terminated, and the vaccination of this dose group or higher dose group will not be carried out, and the study of other dose groups will continue. If this happens at a low dose, the study will be suspended / terminated.

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 18 and 45 years at the first vaccination;
* Be able to understand and comply with the request of the protocol, and sign written informed consent;
* Be able to read, understand and complete diary card;
* According to the medical history and the results of physical examination and laboratory examination, the subjects were judged to be in good health
* Women who agree to use effective contraception throughout the study period；

Exclusion Criteria:

Exclusion criteria of first injection

* History of HPV positive；
* History of drug abuse, alcohol abuse or dependence in the last year；
* History of severe allergy (e.g., anaphylaxis and other significant reaction) to any previous vaccines, or allergy to any of the components of investigational vaccine；
* People with low immune function may be diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, tuberculosis, leukemia, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease or other autoimmune conditions；
* People whose spleen has been removed；
* People received the following immunosuppressive therapy in the past year: radiotherapy, cyclophosphamide, imidazolidine, methotrexate, chemotherapy, cyclosporine, leflunomide, tumor necrosis factor- α Antagonists, monoclonal antibody therapy, intravenous immunoglobulin, anti lymphocyte serum, or other known therapies that interfere with immunity;
* People are receiving systemic corticosteroid therapy, or received two or more courses of high-dose corticosteroids for one week one year before enrollment (nasal inhaled corticosteroids or topical corticosteroids can not be excluded);
* People receiving any immunoglobulin products or blood products within the first 3 months, or planning to receive similar products during the study period;
* Inactivated vaccine was inoculated 14 days before inoculation or attenuated vaccine was inoculated 28 days before inoculation;
* Contraindications of intramuscular injection such as thrombocytopenia or other coagulation disorders;
* Blood donation within the first week or planned during the study period;
* Egg donation was planned during the study period;
* Participating in other experimental clinical studies;
* Have been vaccinated with HPV vaccine on the market or have participated in clinical trials of HPV vaccine;
* Failure to comply with the test procedures or planned relocation during the study;
* Fever occurred within 24 hours before inoculation (axillary temperature > 37 ℃);
* Pregnant women (blood pregnancy test or urine pregnancy test positive) or lactating women;
* There is clinical evidence of purulent cervicitis;
* Having serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension, diabetes and drug uncontrollable;
* Acute infection;
* Other abnormalities, which may confuse the results of the study, or which are not in line with the maximization of the interests of the subjects, can be excluded by the judgment of the investigators.

Exclusion criteria for 2nd or 3rd dose vaccination

* having severe allergic reaction during the first or second dose of vaccination and cannot continue to be vaccinated according to the judgment of investigators;
* The serious adverse reactions with the previous vaccination were related, and the investigators judged that they could not continue to be vaccinated;
* After the first vaccination, the newly discovered or newly occurred serious medical diseases, coagulation dysfunction, etc. can not continue to be vaccinated according to the judgment of the investigators;

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Women Aged 18 to 45 Years
Enrollment: 240 (Estimated)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of local reaction AEs | Up to 7 days following each dose
  Occurrence of local reaction AEs up to 7 days following each dose
Occurrence of systemic AEs | Up to 7 days following each dose
  Occurrence of systemic AEs up to 7 days following each dose
Occurrence of AEs | From dose1 to 30 days after each dose
  Occurrence of AEs from dose1 to 30 days after each dose

SECONDARY OUTCOMES:
Occurrence of SAEs | From dose1 to 30 days after each dose and from dose1 to 12 months after first dose
  Occurrence of SAEs from dose1 to 30 days after each dose and from dose1 to 12 months after first dose
Abnormal hematology and chemistry laboratoty values 3 days after each dose | 3 days after each dose
  Changes in laboratory test indicators (including white blood cell count, lymphocyte count, neutrophils, platelets, hemoglobin, ALT, AST, total bilirubin, fasting blood glucose, creatinine) 3 days after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Guanyun Country CDC, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCormack PL, Joura EA. Quadrivalent human papillomavirus (types 6, 11, 16, 18) recombinant vaccine (Gardasil(R)): a review of its use in the prevention of premalignant genital lesions, genital cancer and genital warts in women. Drugs. 2010 Dec 24;70(18):2449-74. doi: 10.2165/11204920-000000000-00000. PMID 21142263
- [Result] Villa LL, Ault KA, Giuliano AR, Costa RL, Petta CA, Andrade RP, Brown DR, Ferenczy A, Harper DM, Koutsky LA, Kurman RJ, Lehtinen M, Malm C, Olsson SE, Ronnett BM, Skjeldestad FE, Steinwall M, Stoler MH, Wheeler CM, Taddeo FJ, Yu J, Lupinacci L, Railkar R, Marchese R, Esser MT, Bryan J, Jansen KU, Sings HL, Tamms GM, Saah AJ, Barr E. Immunologic responses following administration of a vaccine targeting human papillomavirus Types 6, 11, 16, and 18. Vaccine. 2006 Jul 7;24(27-28):5571-83. doi: 10.1016/j.vaccine.2006.04.068. Epub 2006 May 15. PMID 16753240
- [Result] Palmieri B, Poddighe D, Vadala M, Laurino C, Carnovale C, Clementi E. Severe somatoform and dysautonomic syndromes after HPV vaccination: case series and review of literature. Immunol Res. 2017 Feb;65(1):106-116. doi: 10.1007/s12026-016-8820-z. PMID 27503625